CLINICAL TRIAL: NCT04642989
Title: The Effect of Facial Effleurage on Acute Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017/035
Record Dates: First submitted 2020-05-26; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Rhinosinusitis Acute
Keywords: Osteopathic Manipulative Treatment
MeSH Terms: interventions — Manipulation, Osteopathic; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not informed of the treatment group they are randomized into
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Healthy Control + Sham Treatment (Sham Comparator): Healthy participants who received the sham treatment
  Interventions: Other: Sham Treatment
- Healthy Control + Facial Effleurage (Active Comparator): Healthy participants who received the Facial Effleurage treatment
  Interventions: Other: Facial Effleurage
- Acute Rhinosinusitis + Antibiotics (Active Comparator): Sick participants who received the recommended antibiotics
  Interventions: Drug: Antibiotics
- Acute Rhinosinusitis + Sham Treatment (Sham Comparator): Sick participants who received the sham treatment
  Interventions: Other: Sham Treatment
- Acute Rhinosinusitis + Facial Effleurage (Experimental): Sick participants who received the Facial Effleurage treatment
  Interventions: Other: Facial Effleurage
- Acute Rhinosinusitis + Sham Treatment + Antibiotics (Sham Comparator): Sick participants who received the recommended antibiotics and the sham treatment
  Interventions: Other: Sham Treatment; Drug: Antibiotics
- Acute Rhinosinusitis + Facial Effleurage + Antibiotics (Experimental): Sick participants who received the recommended antibiotics and the Facial Effleurage treatment
  Interventions: Other: Facial Effleurage; Drug: Antibiotics

INTERVENTIONS:
Other: Sham Treatment — All movements of facial effleurage except applying pressure
  Arms: Acute Rhinosinusitis + Sham Treatment; Acute Rhinosinusitis + Sham Treatment + Antibiotics; Healthy Control + Sham Treatment
Other: Facial Effleurage — Facial massage to remove any lymphatic blockages
  Other Names: Osteopathic Manipulative Therapy
  Arms: Acute Rhinosinusitis + Facial Effleurage; Acute Rhinosinusitis + Facial Effleurage + Antibiotics; Healthy Control + Facial Effleurage
Drug: Antibiotics — Appropriate "standard-of-care" antibiotics as determined by the physician.
  Arms: Acute Rhinosinusitis + Antibiotics; Acute Rhinosinusitis + Facial Effleurage + Antibiotics; Acute Rhinosinusitis + Sham Treatment + Antibiotics

SUMMARY:
Rhinosinusitis accounts for 12% of the total antibiotic prescriptions filled in the United States annually; however, the majority of rhinosinusitis cases have been proposed to have a viral etiology, or are capable of spontaneously resolving. This overuse of antibiotics is contributing to the development of antibiotic-resistant human pathogenic bacteria, and increasing patient mortality to previously easily cured diseases. This is also causing an unnecessary financial burden especially for uninsured, rural families. Facial Effleurage (FE) is an osteopathic manipulative therapy that allows physicians an alternative therapy to prescribing antibiotics; however, the only scientific literature on the technique is weak in design and execution. This will be a randomized, placebo-controlled clinical trial to test the ability of FE to reduce symptom severity over time, reduce the cellular infiltrate into the nasal cavity, and to more quickly resolve the symptoms of rhinosinusitis compared to antibiotic treatment. This methodical approach to the efficacy of FE has the potential to impact the treatment recommendations of physicians immediately, and to convince more physicians to prescribe less antibiotics and rely more heavily on FE.

ELIGIBILITY:
Inclusion Criteria:

* Presents with no acute disease OR
* Presents with anterior/posterior mucopurulent drainage and nasal obstruction/facial pain/pressure/fullness
* Independently and without coercion read, understood, and signed the informed consent form
* Is between 18-69 years old.

Exclusion Criteria:

* History of: cancer, HIV, HIV exposure, osteoporosis, acute hepatitis, cystic fibrosis, type-1 diabetes, taking insulin for diabetes, deep vein thrombosis, pulmonary embolism
* History of recent trauma to the liver or spleen or surgery within the past 6 months
* Currently pregnant or nursing
* Have a comorbidity that requires antibiotics or antiviral therapy
* Have a fever greater than 102.5F
* Used topical antimicrobials in the past 30 days
* Taken oral antimicrobials in the past 15 days
* Participated in a clinical trial in the past 6 months
* Have current face or neck bone fractures
* Have abscesses, incisions, or nasal polyps visible on physical examination
* Need to be hospitalized for any reason

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Symptom Severity | 7 days
  SinoNasal Outcome Test-20 questionnaire. The scale is from 0-100 where 0 indicates no symptoms and 100 is the worst symptoms possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Via College of Osteopathic Medicine, Spartanburg, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Any identifying information obtained during the course of this study will be kept confidential. The results of this study, including but not limited to laboratory, clinical, or statistical data may be published. However, no names or other personally identifying information will be published. All subjects participating in this study will be assigned a unique identifier to de-identify their information. The patient number and identifying information will only be on one form during enrollment. All other documents will utilize the patient number. There will be a key that matches each identifier to the study participant. This key will be kept separately from the collected study data and only the study coordinator will have access to it. These records will be kept private in-so-far as permitted by law. All identifiable information will be stored on password-protected computers or in locked file cabinets.